CLINICAL TRIAL: NCT03268356
Title: Clinical Investigation of a Local Osteo-Enhancement Procedure's (LOEP) Ability to Strengthen the Contralateral Femur of Women After a Fragility Fracture of the Hip in Hong Kong
Brief Title: STRONG - Study of AGN1 LOEP for the Treatment of the Contralateral Femur After Fragility Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AgNovos Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PST-HK-100.1
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Hip Fractures; Osteoporosis, Postmenopausal
MeSH Terms: conditions — Hip Fractures; Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AGN1 Treatment (Other): Subjects who have suffered a fragility hip fracture in one hip, sign the consent form and meet the inclusion and none of the exclusion of the study will receive the AGN1 Femoral Local Osteo-Enhancement Procedure (LOEP™) in the non-fractured hip.
  Interventions: Device: AGN1 Femoral Local Osteo-Enhancement Procedure Kit

INTERVENTIONS:
Device: AGN1 Femoral Local Osteo-Enhancement Procedure Kit — A procedure that is intended to replace lost bone and increase the strength of the proximal femur in individuals with osteoporosis of the femoral neck.
  Other Names: AGN1 Femoral LOEP™

SUMMARY:
To evaluate the procedure and safety profile of the AGN1 Femoral LOEP Kit. This pilot study will be used to evaluate AGN1 Femoral LOEP treatment in a contralateral proximal femur during hip fracture repair.

DETAILED DESCRIPTION:
The research will be conducted as a prospective single-center study within Hong Kong. The maximum number of subjects to be treated is twenty (20). This will be a non-randomized and non-blinded study.

Subjects having had a fragility hip fracture on one side will be treated with LOEP in the contralateral non-fractured proximal femur in the same operative session as the surgical repair of the fractured hip. A fragility fracture is defined as a fracture resulting from a fall from standing height.

All subjects will undergo hip fracture repair as recommended by the treating orthopedic surgeon. Repair may include nailing, plates, screws and hip prosthesis.

Subjects may continue to receive, or when appropriate, can be commenced on a treatment regime for osteoporosis. This decision will be made by the treating physician who will determine the best course of action for each patient. The outcome of this decision will have not affect the patient's eligibility for this trial.

Follow-up visits will be conducted at three (3) months, six (6) months, twelve (12) months, and twenty-four (24) months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a postmenopausal female
2. Subject has a low-energy fragility hip fracture in one hip and will undergo surgical repair of the fractured hip.
3. Subject is ≥ 65 years of age.
4. Subject has willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full duration of the study.
5. Subject is capable of giving written informed consent to participate in the study.

Exclusion Criteria:

1. Subject has a prior diagnosis of secondary osteoporosis.
2. Subject has history of any hip surgery or previous hip fracture in the non-fractured hip.
3. Subject has progressive increase in undiagnosed hip pain over the previous six (6) months that in the opinion of the Investigator may suggest other underlying bone or joint pathology (e.g. osteoarthritis, fracture, etc.).
4. Subject has serum calcium levels outside the normal lab range as per local guidelines and reference ranges.
5. Subject has moderate to severe renal insufficiency as per local guidelines and reference ranges.
6. Subject has insulin-dependent diabetes mellitus (IDDM).
7. Subject has Body Mass Index (BMI) > 30.
8. Subject exhibits excessive smokeless tobacco use or excessive smoking as determined by the principal investigator*.
9. Subject exhibits excessive alcohol consumption as determined by the principal investigator*.
10. Subject has radiological evidence of gross bony or joint pathology of the non-fractured hip.
11. Subject treated with corticosteroids or systemic glucocorticoids for ten (10) days in the previous six (6) months.
12. Subject has history of oral or parenteral use of immune-suppressive drugs in the previous twelve months.
13. Subject has history of metabolic bone disease other than osteoporosis (eg. Paget's disease).
14. Subject has a history of auto-immune arthritic diseases including rheumatoid, psoriatic, or those associated with systemic lupus erythematosus, spondyloarthropathy, Reiter's Syndrome or Crohn's Disease.
15. Subject has a history of radiation therapy to the hip or pelvic region.
16. Subject has history of chemotherapy treatment for any condition within the previous five years.
17. Subject has history of any diagnosis and treatment of malignancies (excluding basal cell carcinoma) within the previous five years.
18. Subject has known allergies to implanted device.
19. Subject has severe comorbidity or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate.
20. Subject is currently enrolled in another clinical study.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment or Device Emergent Serious Adverse Events | 24 Months
  Incidence of all serious adverse events (SAEs) occurring from the day of procedure through the twenty-four (24) month follow-up period determined to be definitely related to Femoral LOEP and/or the AGN1 device.

SECONDARY OUTCOMES:
Incidence of Non-Treatment Emergent Fragility Fractures | 24 Months
  Incidence of fragility fractures unrelated to the device or procedure occurring during the follow-up period.
Incidence of Treatment or Device Emergent Adverse Events | 24 Months
  Incidence of all adverse events occurring from the day of procedure through the twenty-four (24) month follow-up determined to be definitely related to Femoral LOEP and/or the AGN1 device.
Change in Bone Mineral Density between Baseline and 12 Months | 12 Months
  Evaluation of bone mineral density (BMD) post-procedure at twelve (12) months.
Change in Bone Mineral Density between Baseline and 24 Months | 24 Months
  Evaluation of bone mineral density (BMD) post-procedure at twenty-four (24) months.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fang, MD, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital - Department of Orthopaedics and Traumatology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website — http://www.agnovos.com